CLINICAL TRIAL: NCT07137832
Title: OPtimizing REperfusion by Intra-Arterial ThRomboLysis as Adjunct to Endovascular Treatment for Medium Vessel Occlusion (PEARL-MeVO): A Multicenter, Prospective, Randomized Controlled, Open-label, Blinded-Endpoint Clinical Trial
Brief Title: OPtimizing REperfusion by Intra-Arterial ThRomboLysis as Adjunct to Endovascular Treatment for Medium Vessel Occlusion
Acronym: PEARL-MeVO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2025-574-02
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intra-arterial thrombolysis as adjunct to endovascular treatment, in addition to standard medical treatment
  Interventions: Combination Product: Intra-arterial thrombolysis as adjunct to endovascular treatment
- Control group (Active Comparator): Only standard medical treatment
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Combination Product: Intra-arterial thrombolysis as adjunct to endovascular treatment — Intra-arterial thrombolysis as adjunct to endovascular treatment, in addition to standard medical treatment
  Arms: Intervention group
Other: Standard medical treatment — Standard medical treatment
  Arms: Control group

SUMMARY:
PEARL-MeVO is an investigator-initiated, multicenter, prospective, randomized controlled, open-label, blinded endpoint (PROBE) clinical trial aiming at evaluating the efficacy and safety of intra-arterial thrombolysis as adjunct to endovascular treatment in improving 90-day functional outcome in acute ischemic stroke patients due to medium vessel occlusion (MeVO) within 24 hours of symptom onset.

DETAILED DESCRIPTION:
PEARL-MeVO is an investigator-initiated, multicenter, prospective, randomized controlled, open-label, blinded endpoint (PROBE) clinical trial aiming at evaluating the efficacy and safety of intra-arterial thrombolysis as adjunct to endovascular treatment in improving 90-day functional outcome in acute ischemic stroke patients due to medium vessel occlusion (MeVO) within 24 hours of symptom onset. The primary outcome is the proportion of patients with a 90-day modified Rankin Scale (mRS) of 0-1. Eligible patients will be randomly assigned at a ratio of 1:1 into the intervention group to receive intra-arterial thrombolysis as adjunct to endovascular treatment, or the control group to receive only standard medical management. A total of 530 participants (265 per group) are anticipated to be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Clinical diagnosis of acute ischemic stroke.
3. CT angiography (CTA) or MR angiography (MRA) confirmed primary isolated medium vessel occlusion (i.e. an occlusion of the co-/non-dominant M2, the M3/M4 segment of the MCA, the A1/A2/A3 segment of the ACA, or the P1/P2/P3 segment of the PCA).
4. Baseline NIHSS ≥6.
5. Treatment (arterial puncture) can be initiated 5.1 Within 6 hours of last known well (LKW) OR 5.2 Within 6 to 24 hours of LKW AND evidence of salvageable brain tissue on CT perfusion or perfusion-diffusion MRI (ischemic core volume <50mL, hypo-perfused tissue volume to ischemic core volume ratio >1.4, mismatch volume >10mL). Hypo-perfused tissue is defined as Tmax >6s on CT perfusion or perfusion MRI. Ischemic core is defined as rCBF <30% on CT perfusion or ADC <620μm2/s on diffusion MRI.
6. Signed informed consent.

Exclusion Criteria:

1. Evidence of intracranial hemorrhage.
2. Pre-stroke mRS score ≥ 2.
3. Rapidly improving symptoms, in the judgment of the managing clinician that the improvement is likely to result in the patient having an NIHSS score of <6 at randomization.
4. The intervention procedure is unlikely to be completed as assessed by the investigator.
5. Suspected cerebral vasculitis, septic embolization, or vascular occlusion due to infective endocarditis.
6. Suspected arterial dissection.
7. Severe allergy to contrast agents (non-mild rash allergy) or absolute contraindication to iodine contrast.
8. Known genetic or acquired bleeding disposition or anticoagulant factors deficiency.
9. Coagulation disorder with INR >1.7 or use of new oral anticoagulants within 48 hours prior to symptom onset.
10. Platelet count <50×10^9/L.
11. Any active or recent bleeding (gastrointestinal, urinary tract bleeding, etc.), or previous parenchymal organ surgery or biopsy in the last 1 month.
12. Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, refractory to treatment.
13. Known severe renal insufficiency with glomerular filtration rate <30 ml/min or blood creatinine >220 μmol/L (2.5 mg/dl).
14. Radiological confirmed evidence of mass effect or intracranial tumour (except small meningioma).
15. Anticipated life expectancy <6 months due to advanced disease (e.g., malignancy, severe cardiopulmonary disease, etc.).
16. Women who are pregnant or breastfeeding.
17. Participation in other clinical trials.
18. Any condition that, in the judgment of the investigator, makes the patient unsuitable for this study or where this study may impose a significant risk to the patient (e.g., inability to understand and/or comply with study procedures and/or follow-up due to psychiatric disorders, cognitive or emotional impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-1 | 90 (±14) days
  The proportion of mRS 0-1 at 90 (±14) days.

SECONDARY OUTCOMES:
Level of disability | 90 (±14) days
  The shift analysis of mRS at 90 (±14) days (mRS 5 and 6 merged)
The modified Rankin Scale score (mRS) 0-2 | 90 (±14) days
  The proportion of mRS 0-2 at 90 (±14) days;
Quality of life (EQ-5D-5L) | 90 (±14) days
  Quality of life measured by the EQ-5D-5L scale score at 90 (±14) days
Neurologic deficit (NIHSS score) changes | 24 (±12) hours
  The change of NIHSS score from baseline at 24 (±12) hours

OTHER OUTCOMES:
Safety outcome: Symptomatic intracranial hemorrhage (sICH) | 24 (±12) hours
  Symptomatic intracranial hemorrhage (sICH) within 36 hours (according to Heidelberg criteria)
Safety outcome: Any intracranial hemorrhage | 24 (±12) hours
  Any intracranial hemorrhage within 36 hours (according to Heidelberg classification);
Safety outcome: Mortality | 90 (±14) days
  All-cause mortality within 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from the Principal Investigator upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the trial completion.
Access Criteria: The IPD will be available from the Principal Investigator upon reasonable request 6 months after the trial completion.